CLINICAL TRIAL: NCT05120180
Title: Postoperative Upper Limb Edema and Dysfunction Generated by Axillary Nodes Excision With or Without Axillary Vein Branches Reservation in Breast Cancer Patients: a Prospective, Multiple-center, Double-blinded, Randomized Controlled Study
Brief Title: Effect of ALND With Vein Branches Reservation on Postoperative Upper Limb Edema and Dysfunction in Breast Cancer
Acronym: PLEDGE-Surgery
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xiangyun Zong (Other)
Responsible Party: Sponsor-Investigator, Xiangyun Zong, Head of Breast Cancer, Principal Investigator, Clinical Professor, Shanghai Jiao Tong University Affiliated Sixth People's Hospital
Organization: Shanghai Jiao Tong University Affiliated Sixth People's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: JTU-6H-20211011001
Record Dates: First submitted 2021-10-25; First posted 2021-11-15 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Breast Cancer Lymphedema
Keywords: Breast Cancer; Axillary Lymph Node Dissection; Post-mastectomy Lymphedema; Upper Limb Dysfunction; Axillary Vein Branches Reservation
MeSH Terms: conditions — Breast Cancer Lymphedema; Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Branches Sparing (Experimental): The patients in this arm will undergo axillary lymph node dissection with preserved axillary vein branches
  Interventions: Procedure: axillary lymph node dissection with vein branches reservation
- None Branches Sparing (Active Comparator): The patients in this arm will undergo axillary lymph node dissection without preserved axillary vein branches
  Interventions: Procedure: axillary lymph node dissection without vein branches reservation

INTERVENTIONS:
Procedure: axillary lymph node dissection with vein branches reservation — Spare the vein branches when ALND being performed
  Arms: Branches Sparing
Procedure: axillary lymph node dissection without vein branches reservation — Don't spare the vein branches when ALND being performed
  Arms: None Branches Sparing

SUMMARY:
The purpose of this study is to compare the effects of axillary lymph node dissection with or without axillary vein branches reservation on the affected upper limb edema and dysfunction in breast cancer patients, and to explore the solutions to prevent the affected upper limb edema and dysfunction after ALND.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-69 years old,
* Regardless of gender,
* Breast masses were diagnosed by histology and pathology, stage II -III.
* Clinical palpation of axillary lymph nodes is positive, or
* Axillary lymph node puncture pathology is positive, or
* The multidisciplinary treatment cooperation group (MDT) recommends axillary lymph node dissection,
* Good physical state score (0-2),
* No severe organ complications,
* No congenital or acquired diseases affecting the normal morphology and functional activities of the upper limbs,
* Informed consent, understanding and compliance with research requirements.

Exclusion Criteria:

* Pregnancy or lactation,
* Inflammatory breast cancer,
* Clinical findings of metastatic lesions,
* Sentinel lymph node biopsy was negative,
* History of upper limb or shoulder, chest, back trauma or surgery,
* Previous history of local radiotherapy,
* History of other tumors,
* Vascular embolic disease,
* Those who are unable to comply with the clinical trial requirements for any reason.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Actual)
Dates: Start 2022-01-03 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2029-04-01 (Estimated)

PRIMARY OUTCOMES:
short-term Incidence of lymphedema | 1-, 6-, and 12-month
  short-term Incidence of upper limb lymphedema on affected side after operation
short-term Incidence of dysfunction | 1-, 6-, and 12-month
  short-term Incidence of upper limb dysfunction on affected side after operation

SECONDARY OUTCOMES:
long-term Incidence of lymphedema | 5 yearsye
  long-term Incidence of upper limb lymphedema on affected side after operation
long-term Incidence of dysfunction | 5 years
  long-term Incidence of upper limb dysfunction on affected side after operation

OTHER OUTCOMES:
TFS | 5 years
  tumor-free survival

CONTACTS AND LOCATIONS:
Overall Officials: XIANGYUN ZONG, M.D., Ph.D.P, Study Chair — Shanghai Jiao Tong University School of Medicine
Locations (3):
- China (3):
  - Shanghai Jiao Tong University Affiliated Sixth People's Hospital, Shanghai, Shanghai Municipality
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Shanghai Fengxian Central Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: No